CLINICAL TRIAL: NCT02018952
Title: Ultrasonography Assessment of Septic Arthritis on Native Joint: a Descriptive, Exploratory, Prospective, Multicentric Trial
Brief Title: Ultrasonography Assessment of Septic Arthritis on Native Joint
Acronym: SEPT'ECHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: RC13_0393
Record Dates: First submitted 2013-12-11; First posted 2013-12-23 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Septic Arthritis
Keywords: Septic arthritis; Ultrasonography; Prognosis parameters
MeSH Terms: conditions — Arthritis, Infectious

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ultrasonography assessment (Other)
  Interventions: Other: Ultrasonography assessment

INTERVENTIONS:
Other: Ultrasonography assessment — All patients will be seen at day 0, day 4, day 15 and at 3 months. These visits are usually programmed. Only monitoring ultrasonography, a non invasive exam, and self-administered questionnaires will be made, additional to standard exams for all patients included (no control group).
  Day 0 :
  * Information of patient and no opposition getting
  * Clinical exam
  * Laboratory tests
  * Radiography of the targeted joint
  * Ultrasonography of the targeted joint and controlateral joint (about 20 minutes)
  Day 4 :
  * Clinical exam
  * Laboratory tests
  * Ultrasonography of the targeted joint and controlateral joint (about 20 minutes)
  Day15 :
  * Clinical exam
  * Laboratory tests
  * Ultrasonography of the targeted joint and controlateral joint (about 20 minutes)
  M3 :
  * Clinical exam
  * Laboratory tests
  * Radiography of the targeted joint
  * Ultrasonography of the targeted joint and controlateral joint (about 20 minutes)
  * Functional outcome

SUMMARY:
The aim of this trial is to study the interest of ultrasonography among patients with septic arthritis.

Currently, ultrasonography is useful for detecting small fluid effusions, for examining otherwise inaccessible joints, such as the hip and for helping the joint aspiration.

Accurate assessment of disease activity and joint damage in septic arthritis is important for monitoring treatment efficiency and for prediction of the outcome of the disease.

Nowadays, magnetic resonance imaging (MRI) provides better resolution than radiography or tomography for the detection of joint effusion and for differentiation between bone and soft tissue infectious. The sensibility is reported to be nearly 100% with a specificity of more than 75%.

However, MRI is expensive and not rapidly accessible.

Therefore, ultrasonography, a non invasive, painless, inexpensive, and non radiating exam can be used to assess the presence and extent of inflammation, destruction, and tissue response.

The objective is to describe, using ultrasonography, the abnormalities joint structure influenced the septic arthritis evolution and prognosis.

The investigators hope, at the end of this study, to evaluate ultrasonography interest in septic arthritis and to establish ultrasonography prognosis factors to predict treatment efficiency and functional outcome.

ELIGIBILITY:
Inclusion Criteria:

* Major patients hospitalized in Rheumatology, Infectiology, Orthopedy Department (hospital of Nantes, of La Roche sur Yon and of Saint-Nazaire) with a septic arthritis of shoulder, or elbow, or wrist , or hip, or knee, or ankle on native joint, with positive microbiologic culture joint fluid or positive hemoculture; the diagnosis was based on positive histology or imagery with an inflammatory joint fluid if the microbiologic cultures (hemoculture or joint effusion) were negative.

Exclusion Criteria:

* Presence of material on the targeted joint
* Age < 18 years old
* Patients under guardianship
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Abnormalities joint structure influencing the septic arthritis evolution and prognosis | 15 months
  Ultrasonography description of :
  * synovium aspect : homogeneous, nodular
  * maximum thickness synovium
  * synovium doppler signal (grade 0, 1, 2, 3)
  * presence and aspect of joint effusion : anechoic, hypo/hyperechoic, heterogeneous
  * presence and aspect of bone erosions : single, minimal/deep, multiple, minimal/ deep
  * presence of a synovium partitioning
  * soft tissue aspect : cellulitis, myelitis

SECONDARY OUTCOMES:
The evolution of the abnormalities joint structure using ultrasonography | 15 months
  To describe the evolution of ultrasonography parameters during the monitoring and to research a link between those ultrasonography parameters and prognostic indicators : ultrasonography parameters at day 0, Day 4, Day 15, and 3 months.
Return delay apyrexia | 15 months
  To describe the evolution of ultrasonography parameters during the monitoring and to research a link between those ultrasonography parameters and prognostic indicators : Return delay apyrexia.
Delay of surgical management | 15 months
  To describe the evolution of ultrasonography parameters during the monitoring and to research a link between those ultrasonography parameters and prognostic indicators : Delay of surgical management.
Normalization of C Reactive Protein levels | 15 months
  To describe the evolution of ultrasonography parameters during the monitoring and to research a link between those ultrasonography parameters and prognostic indicators : Normalization of C Reactive Protein levels.
Measure of range of motion at 3 months | 15 months
Percentage of decreased range of motion relative to normal range of motion at 3 months | 15 months
Pain at rest measured by scale at 3 months | 15 months
Pain during activity measured by scale at 3 months | 15 months
Functional outcome score Short Form (SF) 36 at 3 months | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Benoît LE GOFF, Doctor, Principal Investigator — Nantes University Hospital; Grégoire CORMIER, Doctor, Study Chair — CHD La Roche sur Yon; Oriane MEROT, Doctor, Principal Investigator — CH Saint-Nazaire
Locations (3):
- France (3):
  - CH La Roche-sur-Yon, La Roche-sur-Yon, La Roche-sur-Yon
  - CH Saint-Nazaire, Saint-Nazaire, Saint-Nazaire
  - CH de Nantes, Nantes